CLINICAL TRIAL: NCT04044586
Title: HIV and HCV Infections in 2 Communes From the Battambang Province, Cambodia: Prevalence Rates, Viral Strains, and Unsafe Injection Practices (12352 ANRS ROK INVEST)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University of Health Sciences, Cambodia (Unknown); Hopital Paul Brousse (Other)
Responsible Party: Sponsor
Other Study IDs: ANRS 12352 ROK INVEST
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: HIV Seropositivity; HCV Infection
Keywords: HIV; HCV; outbreak; prevalence
MeSH Terms: conditions — HIV Seropositivity; Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional survey will be conducted prospectively in 2 communes in the Battambang Province, Roka and Prey Khpos commune. The principal objective of the study is to compare HIV and HCV prevalence rates in three groups of subjects as follows:

* Group 1: subjects living in Roka and Ambaeng Thngae villages where most of HIV and HCV cases were identified during the Roka outbreak in 2014-2015
* Group 2: subjects living in the other 4 villages of the Roka commune (Ta Haen I and II, Pou Batdambang, and Chhung Tradak)
* Group 3: subjects living in selected villages from Prey Khpos commune 1,098 eligible residents will be selected using three-stage cluster sampling method. A structure questionnaire will assess the medical injection practices through face-to-face interview. The study will be conducted into two steps. The first step will be a prevalence study to assess HIV and HCV prevalence rates in three groups of subject; Group 1: subjects living in Roka and Ambaeng Thngae villages where most of HIV and HCV cases were identified during the Roka outbreak; Group 2: subjects living in the other 4 villages of the Roka commune (Ta Haen I and II, Pou Batdambang, and Chhung Tradak) and Group 3: subjects living in villages from Prey Khpos commune).The second step will be the phylogenetic study of HIV. The phylogenetic study of HIV will be performed ONLY if HIV prevalence rates among group 2 and/or group 3 is higher or equal to 0.7% (upper limit of confidence interval of HIV prevalence estimated in Cambodia)

DETAILED DESCRIPTION:
Objectives

1. General objective

   The principal objective of the study is to compare HIV and HCV prevalence rates in three groups of subjects as follows:
   * Group 1: subjects living in Roka and Ambaeng Thngae villages where most of HIV and HCV cases were identified during the Roka outbreak in 2014-2015
   * Group 2: subjects living in the other 4 villages of the Roka commune (Ta Haen I and II, Pou Batdambang, and Chhung Tradak)
   * Group 3: subjects living in selected villages from Prey Khpos commune belonging to the Battambang Province.
2. Specific objectives

Given the results we obtained during the investigation of the Roka nosocomial outbreak (2014-15), specific objectives are defined as follows:

* Risk of geographical spread of clustered HCV strains from Roka or Ambaeng Thngae villages to other villages of the Roka commune
* Risk of geographical spread of clustered HIV strains from Roka or Ambaeng Thngae villages to other villages of the Roka commune if the HIV prevalence of Group 2 and/or Group 3 is higher or equal to 0.7% (upper limit of confidence interval of HIV prevalence estimated in Cambodia).
* Comparison of unsafe injection and/or medical practices between the three groups

Methodology This cross-sectional survey will be conducted prospectively in 2 communes in the Battambang Province, i.e. the Roka commune and Prey Khpos commune of the Battambang province. A total of 1,098 eligible residents will be selected according to a three-stage cluster sampling method conducted in the selected sites. A structure questionnaire will assess the medical injection practices through a face-to-face interview. The study will be conducted into two steps. The first step will be a prevalence study to assess HIV and HCV prevalence rates in three groups of subject; Group 1: subjects living in Roka and Ambaeng Thngae villages where most of HIV and HCV cases were identified during the Roka outbreak; Group 2: subjects living in the other 4 villages of the Roka commune (Ta Haen I and II, Pou Batdambang, and Chhung Tradak) and Group 3: subjects living in villages from Prey Khpos commune belonging to the Battambang Province.

The second step will be the phylogenetic study of HIV. The phylogenetic study of HIV will be performed ONLY if HIV prevalence rates among group 2 and/or group 3 is higher or equal to 0.7% (upper limit of confidence interval of HIV prevalence estimated in Cambodia). If the result of HIV prevalence rates among group 2 and group 3 is lower or equal to 0.6% (HIV prevalence estimated in Cambodia), the phylogenetic study of HIV will NOT be performed.

A blood test will be done for HIV and HCV serological antibody screening. For the participants known as HIV positive and/or under ART treatment with NCHADS or as HCV positive, HCV and/or HIV antibody test will not be repeated for these participants and they will be considered as HCV and/or HIV positive. All individuals who will test positive for HCV will be further assessed for viral load measurements. In case of detectable VL results in plasma HCV strains will be amplified, sequenced, and characterized.

In the second step, all individuals who will test positive for HIV will be further assessed for viral load measurements. In case of detectable VL results in plasma or by using whole blood and/or peripheral blood mononuclear cells (PBMCs) in case of undetectable plasma HIV-1 RNA VL results, viral HIV strains will be amplified, sequenced, and characterized.

All tested participants will get a referral slip to retrieve their results (or those from their child) at health care center in the coverage area. Result disclosure will be provided by the doctor (or midwife or nurse) in each center. In case of positive result for at least one virus, we'll advice for the spouse to be tested as well. The same will be suggested for mothers and/or fathers whose child will be identified as infected. The transportation fee for this referral will be offered by the survey.

The total duration of this survey is expected to be 12 months.

Estimated enrollment 1,098 participants

Statistical methods

1. Sample size The formula for two-group comparison was used to calculate the sample size, taking into account the design effect and refusal rate. The minimum sample size of 366 is required per group. Therefore, the total sample size for the 3 groups of subjects in the 2 communes in Battambang will be 1,098 individuals.
2. Sampling strategies A three-stage cluster sampling method will be used to select the eligible participants among residents in the 2 communes in Battambang. This sampling method will be done according to three steps. First, we will select Roka and Prey Khpos Khpos commune in the Battambang province (a commune that looks alike Roka in terms of number of inhabitants is selected). Second, the Simple Random sampling will be used to select 1414 clusters (which are groups) for each group of study population. Third, simple random sampling strategy will be used to select 26 households from each cluster (group) and only one person will be selected per household. The next adjacent household will be used if the person is not present after 3 visits in the first visited household. If more than one person occupies the visited household, one participant will be randomly selected for blood test and face-to-face interview with the research team. If the selected participant is a child, the face-to-face interviews will be done with parent/legal guardian.
3. Data analysis plan

Data analyses will include:

* Description of the participants' demographic characteristics,
* Comparison of HIV and HCV prevalence rates in 3 different groups (subjects living in Roka and Ambaeng Thngae villages of Roka commune, individuals living in the other 4 villages of the Roka commune, and people living in other villages of Prey Khpos commune in the Battambang) using Chi-squared test,
* Comparison of injection history in subjects living in Roka and Ambaeng Thngae villages of Roka versus residents from other villages using Chi-squared test,
* Comparison of viral strains circulating in Roka and Ambaeng Thngae villages of Roka commune versus those present in other villages.

Finally, multiple logistic regression models will be used to assess the independence of variables. All statistical analysis will be performed using STATA version 13.1 software (StataCorp LP, College Station, USA).

Survey timetable Survey start date: Second semester of 2019 Enrolment period: 2 months Subject participation duration: Cross-sectional study Total survey duration: 12 months Estimated survey/trial completion date: Second semester of 2020

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 18 months to 14 years old
* Adult aged ≥ 15 years old
* Informed consent from the participant/parents
* Resident from the selected villages

Exclusion Criteria:

* Children aged less than 18 months

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three groups of subject will be selected: Group 1: subjects living in Roka and Ambaeng Thngae villages where most of HIV and HCV cases were identified during the Roka outbreak; Group 2: subjects living in the other 4 villages of the Roka commune (Ta Haen I and II, Pou Batdambang, and Chhung Tradak) and Group 3: subjects living in villages from Prey Khpos commune belonging to the Battambang Province. The minimum sample size of 366 is required per group. Therefore, the total sample size for the 3 groups of subjects will be 1,098 individuals.
Sampling Method: Probability Sample
Enrollment: 1098 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Determination of HIV and HCV prevalence rates in 2 communes in Battambang province, as well as basic epidemiological risk factors associated with HIV and HCV infections. | July 2019-December 2020
  For the initial screening, ELISA techniques (Murex) will be used for HIV and HCV antibody (Ab) testing. In case of Ab positivity (for HIV and HCV), VL testing will be performed using the Biocentric HIV RNA assay, and the Omunis HCV RNA Viral Load technique.
  In case of detectable (>1,000 copies/ml) HIV and/or HCV VL results or using peripheral blood mononuclear cells (PBMCs) and/or DBS in case of undetectable plasma HIV-1 RNA VL results, viral strains will be amplified and sequenced by Macrogen as follows: C2V3 env region for HIV, and NS5B gene for HCV.
  The phylogenetic analyses will be done for HCV and for HIV using maximum likelihood tree inference and Bayesian evolutionary analyses to obtain temporal information about the date of origin and age of strains (according to 'molecular clock' approaches). Phylogenetic analysis will be performed with the MEGA6 and BEAST softwares.

SECONDARY OUTCOMES:
2/ Phylogenetic characterization of HCV strains circulating in these areas. 3/ Assessment of injection practices among tested subjects enrolled from the 2 studied communes. | July 2019-December 2020
  The survey will assess the knowledge about medical injections practices and beliefs about efficacy of injections among participants using a questionnaire advocated by the WHO and based on previous results described in literature related to injection practices, consists of structured close-ended questions and will include basic demographic, history of medical injections or IV infusions, history of other medical practices as surgery, endoscopy, dental care, assessment of sexual risk behaviors, beliefs about the efficacy of injections and beliefs about the efficacy of parenteral injections. Other exposure factors will be also included in the questionnaire, such as blood transfusion, haemodialysis, tattooing, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Vonthanak SAPHONN, Principal Investigator — University of Health Sciences, Cambodia
Locations (1):
- University of Health Sciences, Phnom Penh, Cambodia